CLINICAL TRIAL: NCT02477254
Title: Long-term Immunogenicity of a Quadrivalent Human Papillomavirus (HPV) Vaccine in Patients With Systemic Lupus Erythematosus: a Case-control Study
Brief Title: Long-term Immunogenicity of a HPV Vaccine in SLE
Status: Completed | Type: Observational
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, consultant, Tuen Mun Hospital
Other Study IDs: NTWC/CREC/15035
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Vaccination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SLE patients: SLE patients who received HPV vaccination
  Interventions: Biological: Vaccination
- Control subjects: Healthy subjects who received HPV vaccination
  Interventions: Biological: Vaccination

INTERVENTIONS:
Biological: Vaccination — A quadrivalent HPV vaccine

SUMMARY:
To study the 5-year immunogenicity against a quadrivalent HPV vaccine in patients with SLE and healthy controls.

DETAILED DESCRIPTION:
Most cases of human papilloma virus (HPV) infection are asymptomatic, transient and resolve without treatment. However, in some individuals, especially those patients who are immunocompromised because of various underlying diseases and those who are receiving long-term immunosuppressive agents, HPV infection is persistent and may result in genital warts, cervical smear abnormalities, cervical intraepithelial neoplasia (CIN) and rarely cervical cancer.

High-risk HPV serotypes are those which are oncogenic and associated with invasive cancers of the cervix and vulva. Examples are the HPV 16 and HPV 18. HPV 16 accounts for almost half of all cervical cancers whereas HPV 18 infection is present in 10-12% of all cervical cancers.

Systemic lupus erythematosus (SLE) patients are at risk of persistent HPV infection. This is because of the immune aberration related to the disease itself and the immunosuppressive state induced by various treatments. One study of 85 SLE patients revealed a 16.5% prevalence of abnormal Pap smears and 12% prevalence of cervical squamous intraepithelial neoplasia (CIN) on routine screening, which was significantly higher than those figures reported in age-matched healthy women (corresponding figures for abnormal Pap smear and CIN were 5.7% and 2%, respectively). Thus, prevention of HPV infection is important in patients with SLE in order to reduce the incidence of CIN lesions and hence invasive cervical cancers in the long run.

The investigators have conducted a case-control study on the safety and immunogenicity of the quadrivalent HPV vaccine, GARDASIL, in 2010. Fifty female SLE patients and 50 age-matched healthy controls were studied. At month 12 after vaccination, the sero-conversion rates of anti-HPV serotypes 6, 11, 16 and 18 in patients and controls were 82%, 89%, 95%, 76% and 98%, 98%, 98%, 80%, respectively. Injection site reaction was the commonest adverse event (AE) (5%), and the incidence of AEs was comparable between patients with SLE and controls.

The investigators plan to study the long-term immunogenicity (durability of the immune response) of the HPV vaccine in the same cohort of patients and controls followed for 5 years. In particular, in patients with SLE, the investigators would like to evaluate the effect of disease flares and ongoing immunosuppressive treatment on the immune response to the HPV serotypes 5 years after vaccination.

ELIGIBILITY:
Inclusion Criteria:

SLE patients

1. Female patients aged 18-35 years
2. Fulfilling the American College of Rheumatology (ACR) criteria for the classification of SLE
3. Having participated in the investigators' original HPV study in 2010
4. Able to give written informed consent

Controls

1. Women aged 18-35 years, matched those of SLE patients recruited
2. No known chronic medical diseases
3. Having participated in our HPV study in 2010

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SLE patients
  1. Female patients aged 18-35 years
  2. Fulfilling the American College of Rheumatology (ACR) criteria for the classification of SLE
  3. Having participated in the investigators' original HPV study in 2010
  4. Able to give written informed consent
  Controls
  1. Women aged 18-35 years, matched those of SLE patients recruited
  2. No known chronic medical diseases
  3. Having participated in our HPV study in 2010
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibodies to HPV serotypes 6,11,16 and 18 | 5 years
  proportion of subjects in each arm who remains sero-converted for each HPV serotype at 5 years after vaccination

SECONDARY OUTCOMES:
Neutralizing antibodies to HPV serotypes 6,11,16 and 18 | 5 years
  the change in anti-HPV titers at 5 years as compared to 12 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, MD, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Ho LY, To CH. Long-term immunogenicity of a quadrivalent human papillomavirus vaccine in systemic lupus erythematosus. Vaccine. 2018 May 31;36(23):3301-3307. doi: 10.1016/j.vaccine.2018.04.056. Epub 2018 Apr 24. PMID 29699792